CLINICAL TRIAL: NCT00843609
Title: International Navigator Hypoglycaemia Study: Evaluation of the Incidence and Duration of Hypoglycaemia Using the Freestyle Navigator® Continuous Glucose Monitoring System
Brief Title: International Navigator Hypoglycaemia Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Karolinska Institutet (Other); Schneider Children's Medical Center, Israel (Other)
Responsible Party: Tadej Battelino, MD,PhD, Professor of pediatrics, UMC Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INHS1
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia
Keywords: diabetes mellitus, type 1; hypoglycemia; continuous glucose monitoring; HbA1c; glycemic variability
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous glucose monitoring (Experimental): Continuously wearing the FreeStyle Navigator continuous glucose monitor, displaying real-time glucose values and sounding alarms
  Interventions: Device: Navigator continuous glucose monitor (Freestyle Navigator®)
- Control (No Intervention): Using SMBG with standard routine instructions

INTERVENTIONS:
Device: Navigator continuous glucose monitor (Freestyle Navigator®) — Continuous use of the Free Style Navigator for monitoring of glycemia in patients with type 1 diabetes with HbA1c below 7.5 %
  Other Names: Free Style Navigator
  Arms: Continuous glucose monitoring

SUMMARY:
The purpose of this study is to determine if the incidence and duration of hypoglycaemia (low blood sugar) is reduced through the use of the FreeStyle Navigator Continuous Glucose Monitoring System in people with Type 1 diabetes mellitus at good glycemic control. The investigators hypothesize that the access to real-time continuous glucose concentration data along with alarms will enable people with type 1 diabetes at reasonable metabolic control to reduce the time spent in hypoglycaemia.

DETAILED DESCRIPTION:
Background:

Real-time continuous glucose monitoring is expected to allow patients to reduce glycaemic fluctuations and to improve their ability to achieve tight glycaemic control without an increase in the incidence or fear of hypoglycaemia through the availability of high fidelity real-time glucose data and alarms throughout the day. As well as in adults, this may be particularly important in both children and adolescents with type 1 diabetes mellitus (T1DM).

Study Overview:

This is a multicentre, prospective, randomised, controlled, intervention study, being conducted at 3 study centres; Ljubljana in Slovenia, Tel Aviv in Israel and Stockholm in Sweden.

The aim is to enroll 100 subjects (50 adult and 50 paediatric), but enrolling up to 120 eligible subjects to allow for dropouts. The subject population will be randomly assigned 50:50 to either the control group or intervention group.

Subjects will be asked to participate for 7 months, consisting of a one-month 'run-in' period on SMBG followed by a 6-month test period. Enrolment will take place within a 16-week period. A blood sample will be taken for centralized baseline measurement of HbA1c. To be included in the study a subject must have an HbA1c level at inclusion below 7.5 % All subjects will undergo a one-month run-in period. Each subject will be given a FreeStyle blood glucose meter and strips to perform self monitoring of blood glucose (SMBG) according to their standard glycaemic management regime, as advised by their health care professional (HCP).

Subjects will then be required to return to the clinic at the end of the run-in period to have another blood sample taken for centralized measurement of HbA1c and to be randomly assigned to Group 1 (intervention) or Group 2 (control) for the next 6-month test period.

Group 1 will be required to use the FreeStyle Navigator CGM to manage their glycaemic control, wearing individual sensors for a series of five day durations, for the next six months.

Group 2 will continue in the study for the next 6 months using SMBG to manage their glycaemic control with the FreeStyle meter and strips provided. Every second week the subject will wear a 'masked' FreeStyle Navigator sensor for 5 days. Subjects will be encouraged to alternate the days that they wear the FreeStyle Navigator sensors, so that data is obtained from days in both the week and weekend.

Subjects will return to the clinic at 3 months and 6 months (after entering the study test-phase) for centralized HbA1c measurement. Subjects (and parents of paediatric subjects) within the intervention group will also be asked to complete a subject satisfaction questionnaire on their experience with the device.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Type 1 diabetes (> 1year since diagnosis)
* CSII or MDI
* HbA1c at inclusion < 7.5 %
* No concomitant diseases that influence metabolic control
* No current use of CGM

Exclusion Criteria:

* Subject has known allergy to medical grade adhesives
* Subject has a medical condition, which in the Investigator's opinion, may compromise patient safety
* Subject is participating in another study of a glucose monitoring device or drug that could affect glucose measurements or glucose management
* Subject is currently using another CGM device or has used real-time continuous glucose monitoring in the previous 4 weeks
* Subject is receiving peritoneal dialysis solutions containing icodextrin
* Female subject who is pregnant or planning to become pregnant within the planned study duration

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Reduction in time spent in hypoglycaemia, defined as continuous glucose <3.5mmol/l (63mg/dl) (with or without symptomatic hypoglycaemia). | 6 months after randomisation

SECONDARY OUTCOMES:
No concomitant rise in HbA1c | 6 months after randomization
Glycaemic variability | 6 months after randomization
Frequency and area under the curve (AUC) of hypoglycaemia | 6 months after randomization
Quality of Life measures (Fear of Hypoglycaemia score and subject satisfaction questionnaire); | 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Battelino, Prof., Principal Investigator — UMC Ljubljana
Locations (3):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- UMC Ljubljana - University Children's Hospital, Ljubljana, Slovenia
- Karolinska Institutet, Stockholm, Sweden